CLINICAL TRIAL: NCT03376984
Title: Nanodiamonds and Antibiotics Modified Gutta-percha (NDGX) for Non-surgical Root Canal Therapy (RCT) Filler Material
Brief Title: Nanodiamond-Gutta Percha Composite Biomaterials for Root Canal Therapy
Acronym: NDGX
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-001308
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Dental Pulp Diseases; Dental Pulp Necrosis; Nerve Root Pain Nec
Keywords: Root Canal Therapy
MeSH Terms: conditions — Dental Pulp Diseases; Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Gutta Percha (Active Comparator): Subjects in both arms of the study will be receiving standard of care RCT and routine follow-up examinations/assessments at 6 months, 1 year, and 2 years post RCT. For all the patients into the control arm of the study, the root canals will be filled with gutta percha (current standard of care), using the vertical condensation obturation technique (standard of care RCT technique).
  Interventions: Device: Gutta Percha
- ND and Amox modified Gutta Percha (Experimental): Subjects in both arms of the study will be receiving standard of care RCT and routine follow-up examinations/assessments at 6 months, 1 year, and 2 years post RCT. The difference between the two arms will be the root canal filler material used. The root canals for the treatment arm of the study will be filled with gutta percha at the apical third, gutta percha modified with nanodiamonds and amoxicillin (NDGX) will be used for the middle and coronal thirds.
  Interventions: Combination Product: ND and AMOX modified Gutta Percha; Device: Gutta Percha

INTERVENTIONS:
Combination Product: ND and AMOX modified Gutta Percha — Gutta percha reinforced and modified with 5 nm diameter nanodiamonds and amoxicillin
  Other Names: NDGX; NDGP; GPX
  Arms: ND and Amox modified Gutta Percha
Device: Gutta Percha — Gutta percha is a device made from coagulated sap of certain tropical trees intended to fill the root canal of a tooth. The gutta percha is softened by heat and inserted into the root canal, where it hardens as it cools. Gutta percha is classified as Class I (general controls).
  Other Names: GP

SUMMARY:
The purpose of this study is to to compare root canal therapy success between two root canal filler materials: 1) gutta percha (GP), 2) gutta percha modified with nanodiamonds and amoxicillin (NDGX). Gutta percha is the current standard root canal filler material used during non-surgical root canal therapy (RCT). Gutta percha modified with nanodiamonds and amoxicillin is an investigational root canal filler material, not yet FDA approved for use as described in this study. The safety and usefulness of NDGX is being tested in this study in comparison to the current standard of care, gutta percha (GP).

DETAILED DESCRIPTION:
This minimal-risk comparison (non-inferiority) study aims to investigate the advantages of Nanodiamond and Amoxicillin modified gutta percha (NDGX) as a root canal filler material for non-surgical root canal therapy. In comparison with the current standard of care, gutta percha (GP), NDGX benefits the patient because NDGX is stronger, may better prevent bacterial reinfection, and potentially reduces complications of non-surgical root canal therapy (RCT) such as tooth fracture, thereby improving overall treatment prognosis. In this study, patients with non-molar teeth needing root canals will be recruited and randomized into two RCT filler material patient groups, with 27 patients with roots filled with the control (GP), and 27 patients with roots filled with NDGX. All patients will be receiving standard of care, and their involvement in our study will only deviate from standard of care in the informed consent process, initial randomization of the root canal filler material, and clinical data collection for research record (already collected in standard of care) from their visits. All patients in the control arm of the study will undergo root canal therapy in which the root canals will be filled with GP. All patients in the NDGX arm of the study will undergo root canal therapy with canals filled with GP in the apical (lower third) end and NDGX in the middle and top thirds of the root canal. In accordance with the standard of care, patients will ideally commit to a total of five visits over a two year period in line with the current standard of care: one pre-treatment consultation appointment, a root canal therapy appointment, a 6 month follow-up appointment, a 1 year follow-up appointment, and a 2 year follow-up appointment. Following standard of care protocol, additional follow-up appointments prior to the 6 month, 1 year, and 2 year follow-up appointments may be required in the event of infection, persistent pain of the root canal following the treatment, and/or at clinician's discretion. Comparison between the control (GP) and NDGX arms of the study will be based upon patient data collected, which will be used to determine clinical "success" derived from reduction and/or absence of a periapical radiolucency and verified with objective and subjective clinical findings such as patient symptoms. Patient data will be categorized by age, weight, gender, and use of other drugs, which may alter the pain assessment and pilot study success indicators.

ELIGIBILITY:
Inclusion Criteria:

* All of the patients must be over 18 years of age and in need of non-surgical RCT treatment during the consultation visit.

Exclusion Criteria:

* Molar teeth
* Osteoporosis medication or i.v. bisphosphonates
* Dental material allergies
* Allergic to penicillin and/or amoxicillin
* Have MD consult/medically compromised/prophylaxis needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Root canal treatment success | 2 years
  Defined as the reduction and/or absence of in periapical radiolucency (PARL) that is verified with objective and subjective clinical findings such as patient symptoms reported (e.g. reported pain levels).

CONTACTS AND LOCATIONS:
Overall Officials: Dean Ho, Ph.D., Principal Investigator — University of California, Los Angeles; Mo K Kang, Ph.D,D.D.S., Principal Investigator — University of California, Los Angeles; Eric C Sung, D.D.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DK, Kim SV, Limansubroto AN, Yen A, Soundia A, Wang CY, Shi W, Hong C, Tetradis S, Kim Y, Park NH, Kang MK, Ho D. Nanodiamond-Gutta Percha Composite Biomaterials for Root Canal Therapy. ACS Nano. 2015 Nov 24;9(11):11490-501. doi: 10.1021/acsnano.5b05718. Epub 2015 Oct 15. PMID 26452304
- [Background] Lee DK, Kee T, Liang Z, Hsiou D, Miya D, Wu B, Osawa E, Chow EK, Sung EC, Kang MK, Ho D. Clinical validation of a nanodiamond-embedded thermoplastic biomaterial. Proc Natl Acad Sci U S A. 2017 Nov 7;114(45):E9445-E9454. doi: 10.1073/pnas.1711924114. Epub 2017 Oct 23. PMID 29078364